CLINICAL TRIAL: NCT02308293
Title: The Effect of Exercise-induced Hyperlacticacidemia on Counterregulatory Responses, Symptoms, Cognitive Function and Brain Lactate Accumulation During Hypoglycemia in (Hypoglycemic Unaware)Type I Diabetes Patients and Normal Controls
Brief Title: The Role of Endogenous Lactate in Brain Preservation and Counterregulatory Defenses Against Hypoglycemia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Radboud University Medical Center (Other)
Collaborators: Dutch Diabetes Research Foundation (Other); European Foundation for the Study of Diabetes (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: End_lac_sympt
Record Dates: First submitted 2014-11-14; First posted 2014-12-04 (Estimated); Last update posted 2016-11-25 (Estimated); Status verified 2016-04

CONDITIONS: Type 1 Diabetes Mellitus; Hypoglycemia Unawareness
Keywords: Type 1 Diabetes Mellitus; Hypoglycemia unawareness; Lactate; high intensity interval exercise; MRS
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — High-Intensity Interval Training

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- High intensity exercise (Experimental): Subjects will preform a high intensity training exercise (3* 30 seconds all out sprint on a cycle ergometer) to raise plasma lactate levels
  Interventions: Behavioral: High intensity exercise
- Lay down comfortably (Sham Comparator): As a control conditions, subjects wil lay down comfortably and rest
  Interventions: Behavioral: Lay down comfortably

INTERVENTIONS:
Behavioral: High intensity exercise — 3x30 seconds 'all out' sprints
  Arms: High intensity exercise
Behavioral: Lay down comfortably — rest
  Arms: Lay down comfortably

SUMMARY:
Iatrogenic hypoglycemia is the most frequent acute complication of insulin therapy in people with type 1 diabetes (T1DM). Recurrent hypoglycemic events initiate a process of habituation, characterized by suppression of hypoglycemic symptoms, eventually leading to hypoglycemia unawareness, which creates a particularly high risk of severe hypoglycemia. Recent evidence suggest a pivotal role for (brain) lactate in the pathogenesis of hypoglycemia unawareness. Indeed, exogenous lactate administration may preserve brain function and attenuate counterregulatory responses to and symptomatic awareness of hypoglycemia. It is unknown whether endogenous elevation of plasma lactate produces the same effects and whether such effects differ between patients with T1DM with and without hypoglycemia unawareness and healthy controls.

Objective: To investigate the effect of elevated levels of endogenous lactate on brain lactate accumulation and on counterregulatory responses to, symptomatic awareness of and cognitive function during hypoglycemia in patients with T1DM with and without hypoglycemia unawareness and normal controls.

Hypothesis: The investigators hypothesize first that endogenous lactate, when raised through high intensity exercise, preserves neuronal metabolism during subsequent hypoglycemia, which in turn will attenuate counterregulatory hormone responses, appearance of symptoms and deterioration of cognitive function. Second, the investigators posit that these effects will be augmented in patients with hypoglycemia unawareness compared to healthy subjects and T1DM patients with normal awareness as a consequence of greater transport capacity of lactate into the brain.

ELIGIBILITY:
Inclusion criteria for healthy subjects

* Age: 18-40 years
* Body-Mass Index: 18-30 kg/m2
* Blood pressure: <160/90 mmHg
* Recreationally active: i.e. taking part in competitive sport or regular exercise training, of a non-professional nature, once or more a week.

Inclusion criteria T1DM patients with normal hypoglycemic awareness

* Diabetes duration ≥ 1 year
* Age: 18-40 years
* Body-Mass Index: 18-30 kg/m2
* HbA1c: 42-75 mmol/mol (6-9%)
* Outcome Clarke questionnaire: 0-1
* Blood pressure: <160/90 mmHg
* Recreationally active: i.e. taking part in competitive sport or regular exercise training, of a non-professional nature, once or more a week

Inclusion criteria T1DM patients with hypoglycemia unawareness

* Diabetes duration ≥ 1 year
* Age: 18-40 years
* Body-Mass Index: 18-30 kg/m2
* HbA1c: 42-75 mmol/mol (6-9%)
* Outcome Clarke questionnaire: =>3
* Blood pressure: <160/90 mmHg
* Recreationally active

Exclusion criteria:

* Inability to provide informed consent
* Presence of any medical condition that might interfere with the study protocol, such as brain injuries, epilepsy, a major cardiovascular disease event or anxiety disorders
* Use of any medication, except for oral contraceptives
* MR(I) contraindications (pregnancy, severe claustrophobia, metal parts in body)
* Orthopedic and/or neurological diseases that impair exercise
* Cardiopulmonary disease as stated in the 2001 American heart association and 2002 American college of cardiology/American heart association guidelines

Additional exclusion criteria for all T1DM patients:

* Use of any other medication than insulin, except for oral contraceptives or stable thyroxine supplementation therapy
* complications of T1DM, including proliferative retinopathy, neuropathy or nephropathy

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2015-01; Primary Completion 2016-05 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Plasma level of adrenaline in response to hypoglycemia (Adrenaline, measured in arterial plasma) | during 60 m of hypoglycemia

SECONDARY OUTCOMES:
Plasma levels of other counter-regulatory hormones (Levels of counter-regulatory hormones measured in arterial plasma) | During 60 min hypoglycemia
  Levels of counter-regulatory hormones measured in arterial plasma
Glucose infusion rate (Amount of glucose 20% necessary to maintain plasma glucose at steady state values) | During 60 min hypoglycemia
  Amount of glucose 20% necessary to maintain plasma glucose at steady state values
Plasma lactate levels (Lactate levels measured in arterial plasma) | During 60 min hypoglycemia
  Lactate levels measured in arterial plasma
Cognitive functioning, as measured by cognitive tests | During 60 min hypoglycemia
  Cognitive test will be: Dutch State Trait Anxiety Inventory, Digit Span, Stroop color word test, word fluency test, trail making test and Pasat
Plasma levels of inflammatory markers (levels of cytokines) | During 60 min hypoglycemia
  levels of cytokines
Brain perfusion measured with ASL-MRI | During 60 min hypoglycemia
  Brain perfusion measured with ASL-MRI
Brain lactate accumulation measured with 1H-MRS | During 60 min of hypoglycemia
  Brain lactate levels measured with 1H-MRS

OTHER OUTCOMES:
Plasma glucose concentration | During 60 min hypoglycemia
  Plasma glucose concentration, necessary to adjust glucose infusion rate
Plasma insulin concentration (Insulin levels, measured in arterial plasma) | During 60 min hypoglycemia
  Insulin levels, measured in arterial plasma

CONTACTS AND LOCATIONS:
Overall Officials: Bastiaan de Galan, Dr., Principal Investigator — Radboud University Medical Center
Locations (1):
- Radboud umc, Nijmegen, Netherlands

REFERENCES:
- [Background] van de Ven KC, van der Graaf M, Tack CJ, Klomp DW, Heerschap A, de Galan BE. Optimized [1-(13)C]glucose infusion protocol for 13C magnetic resonance spectroscopy at 3T of human brain glucose metabolism under euglycemic and hypoglycemic conditions. J Neurosci Methods. 2010 Jan 30;186(1):68-71. doi: 10.1016/j.jneumeth.2009.10.025. Epub 2009 Nov 11. PMID 19913052
- [Background] van de Ven KC, de Galan BE, van der Graaf M, Shestov AA, Henry PG, Tack CJ, Heerschap A. Effect of acute hypoglycemia on human cerebral glucose metabolism measured by (1)(3)C magnetic resonance spectroscopy. Diabetes. 2011 May;60(5):1467-73. doi: 10.2337/db10-1592. Epub 2011 Apr 4. PMID 21464446
- [Background] van de Ven KC, van der Graaf M, Tack CJ, Heerschap A, de Galan BE. Steady-state brain glucose concentrations during hypoglycemia in healthy humans and patients with type 1 diabetes. Diabetes. 2012 Aug;61(8):1974-7. doi: 10.2337/db11-1778. Epub 2012 Jun 11. PMID 22688331
- [Background] De Feyter HM, Mason GF, Shulman GI, Rothman DL, Petersen KF. Increased brain lactate concentrations without increased lactate oxidation during hypoglycemia in type 1 diabetic individuals. Diabetes. 2013 Sep;62(9):3075-80. doi: 10.2337/db13-0313. Epub 2013 May 28. PMID 23715622
- [Background] Maddock RJ, Casazza GA, Buonocore MH, Tanase C. Vigorous exercise increases brain lactate and Glx (glutamate+glutamine): a dynamic 1H-MRS study. Neuroimage. 2011 Aug 15;57(4):1324-30. doi: 10.1016/j.neuroimage.2011.05.048. Epub 2011 May 27. PMID 21640838
- [Derived] Wiegers EC, Rooijackers HM, van Asten JJA, Tack CJ, Heerschap A, de Galan BE, van der Graaf M. Elevated brain glutamate levels in type 1 diabetes: correlations with glycaemic control and age of disease onset but not with hypoglycaemia awareness status. Diabetologia. 2019 Jun;62(6):1065-1073. doi: 10.1007/s00125-019-4862-9. Epub 2019 Apr 19. PMID 31001674
- [Derived] Wiegers EC, Rooijackers HM, Tack CJ, Groenewoud HJMM, Heerschap A, de Galan BE, van der Graaf M. Effect of Exercise-Induced Lactate Elevation on Brain Lactate Levels During Hypoglycemia in Patients With Type 1 Diabetes and Impaired Awareness of Hypoglycemia. Diabetes. 2017 Dec;66(12):3105-3110. doi: 10.2337/db17-0794. Epub 2017 Sep 21. PMID 28935628
- [Derived] Rooijackers HM, Wiegers EC, van der Graaf M, Thijssen DH, Kessels RPC, Tack CJ, de Galan BE. A Single Bout of High-Intensity Interval Training Reduces Awareness of Subsequent Hypoglycemia in Patients With Type 1 Diabetes. Diabetes. 2017 Jul;66(7):1990-1998. doi: 10.2337/db16-1535. Epub 2017 Apr 18. PMID 28420673